CLINICAL TRIAL: NCT02948660
Title: EEG Dynamics Induced by Zolpidem Forecasts Consciousness Evolution in Prolonged Disorders of Consciousness and Quantification of EEG Reactivity Predicts Recovery of Consciousness
Brief Title: A Promising Tool for Predicting Consciousness Evolution in Prolonged Disorders of Consciousness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Guangzhou University of Chinese Medicine (Other); University of Melbourne (Other); Tianjin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 81571262
Record Dates: First submitted 2016-10-23; First posted 2016-10-28 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-03

CONDITIONS: Disorder of Consciousness
Keywords: Prolonged disorders of consciousness; Zolpidem; EEG; Prognosis; Unresponsive wakefulness syndrome; Minimally conscious state
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with prolonged disorders of consciousness (Experimental): 1. age ≥ 18 years;
  2. presence of unresponsive wakefulness syndrome (UWS) or minimally conscious state (MCS) on admission;
  3. time since onset > 4 weeks;
  4. no history of neurodegenerative or psychiatric diseases.
  All patients were administered 10 mg of zolpidem tartrate tablets via a feeding tube and received EEG-reactivity test.
  Interventions: Drug: Zolpidem Tartrate Tablets
- Healthy volunteers (Experimental): Healthy volunteers without any history of autonomic or any other nervous system disorder were included in this study. They were administered 10 mg of zolpidem tartrate tablets orally.
  Interventions: Drug: Zolpidem Tartrate Tablets

INTERVENTIONS:
Drug: Zolpidem Tartrate Tablets — All participants were administered 10 mg of zolpidem tartrate tablets either via a feeding tube (for patients with prolonged disorders of consciousness) or orally.

SUMMARY:
The research contains two parts. Part 1: To explore whether EEG responses to zolpidem can assess consciousness circuit integrity and predict the evolution of consciousness in patients with prolonged disorders of consciousness; Part 2: To explore if quantitative EEG reactivity might predict the prognosis of disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* presence of unresponsive wakefulness syndrome (UWS) or minimally conscious state (MCS) on admission;
* time since onset > 4 weeks;
* no history of neurodegenerative or psychiatric diseases.

Exclusion Criteria:

* allergic to zolpidem;
* currently receiving zolpidem or related benzodiazepines;
* diagnosed with seizure or status epilepticus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The Coma Recovery Scale-Revised | Six months after enrollment
  The consciousness was independently assessed using CRS-R six months after enrollment by a trained neurologist blinded to the clinical data. Patients who transitioned from UWS to MCS (UWS-MCS) or to emergence from MCS (EMCS) (UWS-EMCS), from MCS minus to MCS plus (MCS--MCS+) or to EMCS (MCS--EMCS), and from MCS to EMCS (MCS-EMCS) were categorized in the improved consciousness group. The unimproved consciousness was defined as a reduced or unchanged level of consciousness at six months.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, doctor, Study Director — Department of Neurology, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Neurology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China